CLINICAL TRIAL: NCT00029146
Title: Carotid Occlusion Surgery Study
Acronym: COSS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pre-specified futility boundary was reached.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Washington University School of Medicine (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, William Powers, Professor of Neurology, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS042167; R01NS041895 (Other Grant/Funding Number: NINDS)
Record Dates: First submitted 2002-01-08; First posted 2002-01-09 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Stroke; Ischemic Attack, Transient; Cerebral Infarction
Keywords: stroke; transient ischemic attack (TIA); carotid arteries; cerebral infarction
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Cerebral Infarction | interventions — Cerebral Revascularization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical group (Experimental): Assigned to undergo extracranial-intracranial arterial bypass in addition to best current practice medical therapy
  Interventions: Procedure: extracranial-intracranial bypass surgery
- Non-surgical group (Active Comparator): Receives best current practice medical therapy
  Interventions: Drug: best medical therapy

INTERVENTIONS:
Procedure: extracranial-intracranial bypass surgery — Surgical anastomosis of a superficial temporal artery branch to a middle cerebral artery branch through a small craniectomy plus best current practice medical therapy
  Other Names: EC-IC Arterial Bypass; STA-MCA Bypass
  Arms: Surgical group
Drug: best medical therapy — best current practice medical therapy
  Arms: Non-surgical group

SUMMARY:
The purpose of this study is to determine if extracranial-intracranial bypass surgery when added to best medical therapy can reduce the subsequent risk of ipsilateral stroke in high-risk patients with recently symptomatic carotid occlusion and increased cerebral oxygen extraction fraction measured by positron emission tomography (PET).

DETAILED DESCRIPTION:
The overall purpose of this research is to determine if a surgical operation called "Extracranial-Intracranial Bypass" can reduce the chance of a subsequent stroke in someone who has complete blockage in one main artery in the neck (the carotid artery) that supplies blood to the brain and has already suffered a small stroke. This surgery involves taking an artery from the scalp outside the skull, making a small hole in the skull and then connecting the scalp artery to a brain artery inside the skull. In this way the blockage of the carotid artery in the neck is bypassed and more blood can flow to the brain. In some people natural bypass arteries develop and the brain is already getting plenty of blood. These people have a low risk of stroke if they take medicine. In other people, no natural bypass arteries develop so less blood flows to their brains. This second group has a much higher risk of stroke while taking medicine, as high as 25-50% within the next two years. It is this second group of people who may benefit from having the bypass operation and who are the candidates for this study.

This bypass surgery is considered experimental because it is not generally performed for this condition and it is unknown whether it leads to a decrease, an increase or no change in the risk of stroke. In order to determine if people fit into this second group of people who may benefit from the bypass operation they need to have a test called a PET scan. The PET scan measures the amount of blood that is getting to the brain and the amount of oxygen that the brain is using. The PET scan uses radioactive oxygen and water and is experimental (not approved by the United States Food and Drug Administration). If the PET scan shows that less blood is getting to the brain, there will be a 50-50 chance (like a coin toss) of receiving the bypass surgery or not. There will then be follow-up visits to the clinic one month later and then every three months for two years to check on the appropriate medical treatment that everyone will receive and to determine who has had a stroke.

The study hypothesis is that extracranial-intracranial bypass surgery when added to best medical therapy can reduce by 40 percent subsequent stroke within two years in participants with recent TIA ('ministroke") or stroke (</= 120 days) due to blockage of the carotid artery and reduced blood flow to the brain measured by PET.

ELIGIBILITY:
Inclusion Criteria:

* Vascular imaging demonstrating occlusion of one or both internal carotid arteries.
* Transient ischemic attack (TIA) or ischemic stroke in the hemispheric carotid territory of one occluded carotid artery.
* Most recent qualifying TIA or stroke occurring within 120 days prior to projected performance date of PET.
* Modified Barthel Index > 12/20 (60/100).
* Language comprehension intact, motor aphasia mild or absent.
* Age 18-85 inclusive.
* Competent to give informed consent.
* Legally an adult.
* Geographically accessible and reliable for follow-up.

Exclusion Criteria:

* Non-atherosclerotic carotid vascular disease. Blood dyscrasias: Polycythemia vera ,essential thrombocytosis, sickle cell disease (SS or SC).
* Known heart disease likely to cause cerebral ischemia (echocardiography not required). This includes the following conditions ONLY: Prosthetic valve, Infective endocarditis, Left atrial or ventricular thrombus, Sick sinus syndrome, Myxoma, Cardiomyopathy with ejection fraction <25%. This is an all-inclusive list. The following conditions are NOT EXCLUSIONS: Atrial fibrillation, patent foramen ovale, atrial septal aneurysm.
* Other non-atherosclerotic condition likely to cause focal cerebral ischemia.
* Any condition likely to lead to death within 2 years.
* Other neurological disease that would confound follow-up assessment.
* Pregnancy.
* Subsequent cerebrovascular surgery planned which might alter cerebral hemodynamics.
* Any condition which in the participating surgeon's judgment makes the subject an unsuitable surgical candidate.
* Participation in any other experimental treatment trial.
* Participation within the previous 12 months in any experimental study that included exposure to ionizing radiation.
* Acute, progressing or unstable neurological deficit. Neurological deficit must be stable for 72 hours prior to the performance of PET.
* If supplemental arteriography is required, allergy to iodine or x-ray contrast media, serum creatinine > 3.0 mg/dl or other contraindication to arteriography.
* If aspirin is to be used as antithrombotic therapy in the perioperative period, those with allergy or contraindication to aspirin are ineligible.
* Medical indication for treatment with anticoagulant drugs, ticlopidine, clopidogrel or other antithrombotic medications such that these medications cannot be replaced with aspirin in the perioperative period as deemed necessary by the COSS neurosurgeon if the participant is randomized to surgical treatment.
* Remediable medical conditions. Patients with the following conditions can become eligible if the exclusion criterion no longer applies within 120 days of onset of the most recent qualifying event: Uncontrolled diabetes mellitus (FBS > 300 mg%/16.7 mmol/L), Uncontrolled hypertension (systolic BP>180, diastolic BP >110), Unstable angina, Uncontrolled hypotension (diastolic BP < 65).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2002-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Powers, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Grubb RL Jr, Derdeyn CP, Fritsch SM, Carpenter DA, Yundt KD, Videen TO, Spitznagel EL, Powers WJ. Importance of hemodynamic factors in the prognosis of symptomatic carotid occlusion. JAMA. 1998 Sep 23-30;280(12):1055-60. doi: 10.1001/jama.280.12.1055. PMID 9757852
- [Background] Derdeyn CP, Gage BF, Grubb RL Jr, Powers WJ. Cost-effectiveness analysis of therapy for symptomatic carotid occlusion: PET screening before selective extracranial-to-intracranial bypass versus medical treatment. J Nucl Med. 2000 May;41(5):800-7. PMID 10809195
- [Background] Adams HP Jr, Powers WJ, Grubb RL Jr, Clarke WR, Woolson RF. Preview of a new trial of extracranial-to-intracranial arterial anastomosis: the carotid occlusion surgery study. Neurosurg Clin N Am. 2001 Jul;12(3):613-24, ix-x. PMID 11390318
- [Background] Grubb RL Jr, Powers WJ, Derdeyn CP, Adams HP Jr, Clarke WR. The Carotid Occlusion Surgery Study. Neurosurg Focus. 2003 Mar 15;14(3):e9. doi: 10.3171/foc.2003.14.3.10. PMID 15709726
- [Derived] Grubb RL Jr, Powers WJ, Clarke WR, Videen TO, Adams HP Jr, Derdeyn CP; Carotid Occlusion Surgery Study Investigators. Surgical results of the Carotid Occlusion Surgery Study. J Neurosurg. 2013 Jan;118(1):25-33. doi: 10.3171/2012.9.JNS12551. Epub 2012 Oct 26. PMID 23101451
- [Derived] Powers WJ, Clarke WR, Grubb RL Jr, Videen TO, Adams HP Jr, Derdeyn CP; COSS Investigators. Extracranial-intracranial bypass surgery for stroke prevention in hemodynamic cerebral ischemia: the Carotid Occlusion Surgery Study randomized trial. JAMA. 2011 Nov 9;306(18):1983-92. doi: 10.1001/jama.2011.1610. PMID 22068990

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgical Group | Non-surgical Group
Started | 97 | 98
Completed | 95 | 97
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgical Group | Non-surgical Group | Total
Number analyzed (Participants) | 97 | 98 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 71 | 147
  >=65 years | 21 | 27 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (9) | 58 (9) | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 37 | 65
  Male | 69 | 61 | 130
Region of Enrollment [Number; unit: participants]
  United States | 93 | 94 | 187
  Canada | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Surgical Group:Ipsilateral Ischemic Stroke in 2 Yrs From Randomization and All Stroke & Death Through 30d Post-surgery; Non-surgical Group:Ipsilateral Ischemic Stroke in 2 Yrs From Randomization and All Stroke & Death Through 30d Post-randomization
Description: 2 yr Kaplan-Meier estimates of the proportions.Proportions expressed as percentages for reporting purposes. Ipsilateral ischemic stroke is defined as the clinical diagnosis of a focal neurological deficit due to cerebral ischemia clinically localizable within the internal carotid artery territory distally to the symptomatic occluded internal carotid artery that lasts for more than 24 hours. All stroke is defined as the clinical diagnosis of a focal deficit due to ischemia or hemorrhage clinically localizable to the brain that lasts for more than 24 hours. Death is of any cause.
Time Frame: within 2 yrs of randomization
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
percentage of participants | 21.0 [12.8 to 29.2] | 22.7 [13.9 to 31.6]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; Rates for each group were based on product limit estimates of 2-year rates and their standard errors. The test statistic was calculated as the difference in estimated rates divided by the standard error of that difference. The 2-sided z-statistic was compared to a standard unit normal distribution.The study was terminated early for futility after 195 of the planned 372 participants were enrolled; Test type: Superiority or Other; p = 0.78, 2-sided z-statistic; The difference in estimated rates divided by the standard error of that difference was compared to a standard unit normal distribution; Difference in estimated 2 yr rates = 1.7, 95% CI [-10.4 to 13.8] — Positive indicates lower rate in surgical group

2. Secondary Outcome: All Stroke
Description: 2 yr Kaplan-Meier estimates of the proportions. All stroke is defined as the clinical diagnosis of a focal deficit due to ischemia or hemorrhage clinically localizable to the brain that lasts for more than 24 hours
Time Frame: within 2 yrs of randomization
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
percentage of participants | 23.4 [14.8 to 32.0] | 26.9 [17.6 to 36.2]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; Rates for each group were based on product limit estimates of 2-year rates and their standard errors; Test type: Superiority or Other; p = 0.59, 2-sided z-statistic; [statistical method as in outcome 1, analysis 1]; Difference in estimated 2 yr rates = 3.5, 95% CI 2-sided [-9.2 to 16.1] — Positive indicates lower rate in surgical group

3. Secondary Outcome: Disabling Stroke
Description: 2 yr Kaplan-Meier estimates of the proportions. Disabling stroke is defined as a modified Barthel Index of <12/20 at the first scheduled return visit more than 3 months after the stroke occurred
Time Frame: within two years after randomization
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
percentage of participants | 5.9 [0.8 to 10.4] | 2.4 [0 to 5.6]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; Rates for each group were based on product limit estimates of 2-year rates and their standard errors. The test statistic was calculated as the difference in estimated rates divided by the standard error of that difference; Test type: Superiority or Other; p = 0.27, 2-sided z-statistic; [statistical method as in outcome 1, analysis 1]; Difference in estimated 2 yr rates = -3.2, 95% CI 2-sided [-9.0 to 2.6] — Negative indicates lower rate in non-surgical group

4. Secondary Outcome: Fatal Stroke
Description: 2 yr Kaplan-Meier estimates of the proportions. Fatal stroke is a stroke that in the investigator's opinion led directly to the participants death within 30 days of occurrence
Time Frame: within 2 years after randomization
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
percentage of participants | 1.0 [0 to 3.1] | 2.4 [0 to 5.6]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.50, 2-sided z-statistic; [statistical method as in outcome 1, analysis 1]; Difference in estimated 2 yr rates = 1.3, 95% CI 2-sided [-2.5 to 5.2] — Positive indicates lower rate in surgical group

5. Secondary Outcome: Death
Description: 2 yr Kaplan-Meier estimates of the proportions. Death of any cause
Time Frame: within 2 years after randomization
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
percentage of participants | 1.0 [0 to 3.1] | 5.1 [0.2 to 9.9]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.13, 2-sided z-statistic; [statistical method as in outcome 1, analysis 1]; Difference in estimated 2 yr rates = 4.0, 95% CI 2-sided [-1.2 to 9.7] — Positive indicates lower rate in surgical group

6. Post Hoc Outcome: Any Stroke or Death
Description: 2 yr Kaplan-Meier estimates of the proportions. Any stroke is defined as the clinical diagnosis of a focal deficit due to ischemia or hemorrhage clinically localizable to the brain that lasts for more than 24 hours. Death is of any cause.
Time Frame: within 2 years after randomization
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
percentage of participants | 23.4 [14.8 to 32.0] | 29.9 [20.1 to 39.8]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = .33, 2-sided z-statistic; [statistical method as in outcome 1, analysis 1]; Difference in estimated 2 yr rates = 6.5, 95% CI 2-sided [-6.5 to 19.6] — Positive indicates lower rate in surgical group

7. Secondary Outcome: Modified Rankin 0-1
Description: Proportion with modified Rankin score, dichotomized 0 or 1 vs 2-6.The modifed Rankin (0-6) describes the degree of functional disability. A lower score indicates less functional disability.
Time Frame: at 2 years after randomization or end of trial. Worst case imputed for death and missing values
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
percentage of participants | 49.5 [39.5 to 59.4] | 42.9 [33.1 to 52.7]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; Test type: Superiority or Other; p = 0.41, Fisher Exact; Difference in estimated 2 yr rates = -6.6, 95% CI 2-sided [-20.6 to 7.3] — Negative indicates lower rate in non-surgical group. In this case, lower rate is worse since Rankin 0-1 indicates a good outcome

8. Secondary Outcome: Modified Rankin 0-2
Description: Proportion with Modified Rankin score at 2 yrs, dichotomized 0-2 vs 3-6. The modifed Rankin (0-6) describes the degree of functional disability. A lower score indicates less functional disability.
Time Frame: at 2 years after randomization or end of trial. Worst case imputed for death and missing values
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
percentage of participants | 70.1 [61.0 to 79.2] | 74.5 [65.9 to 83.1]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; Test type: Superiority or Other; p = 0.70, Fisher Exact; Difference in estimated 2 yr rates = 4.4, 95% CI 2-sided [-8.2 to 16.9] — Positive indicates lower rate in surgical group In this case, lower rate is worse since Rankin 0-2 indicates a good outcome

9. Secondary Outcome: Modified Barthel Index 19-20
Description: Modified Barthel Index dichotomized 19-20 vs <= 18. The modifed Barthel Index(0-20) describes the degree of independence in day-to-day self-care activities. A higher score indicates greater independence.
Time Frame: at 2 years after randomization or end of trial. Worst case imputed for death and missing values
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
percentage of participants | 70.1 | 71.4
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; Test type: Superiority or Other; p = 0.85, Fisher's Exact Test

10. Secondary Outcome: Summary SS-QOL Score
Description: Summary Stroke Specific Quality of Life score (1-4) askes how self-reported overall quality of life compares with with that before stroke. A higher score indicates is better.
Time Frame: at 2 years after randomization or end of trial. Worst case imputed for death and missing values
Population: Intention to treat principle.All participants analyzed in the group to which they were originally randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 97 | 98
units on a scale | 3.82 [3.60 to 4.04] | 3.58 [3.37 to 3.79]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; Test type: Superiority or Other; p = 0.13, t-test, 2 sided; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.54 to 0.07] — Negative indicates lower score in non-surgical group.A higher score indicates better quality of life

11. Secondary Outcome: Ipsilateral Ischemic Stroke in 2 Yrs From Randomization and All Stroke & Death Through 30d Post-surgery; Non-surgical Group:Ipsilateral Ischemic Stroke in 2 Yrs From Randomization and All Stroke & Death Through 30d Post-randomization
Description: as for outcome 1
Time Frame: within 2 years of randomization
Population: On-treatment analysis removing four participants assigned to the surgical group who never underwent surgery and censoring on the day of surgery three participants assigned to the nonsurgical group who underwent EC-IC bypass surgery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 93 | 98
percentage of participants | 20.8 [12.4 to 29.1] | 22.3 [13.3 to 31.2]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.81, 2-sided z-statistic; [statistical method as in outcome 1, analysis 1]; Difference in estimated 2 yr rates = 1.5, 95% CI 2-sided [-10.7 to 13.7]

12. Other Pre Specified Outcome: Any Stroke or Death Within 30 Days After Surgery
Time Frame: within 30 days after surgery
Population: Intention-to-treat. All assigned to undergo extracranial-intracranial arterial bypass in addition to best current practice medical therapy
Measure: Number; unit: participants
Arm/Group | Surgical Group
Number analyzed (Participants) | 97
participants | 14

ADVERSE EVENTS:
Time Frame: Surgical group: Within 30 days after surgery for 93 operated and within 30 days after randomization for 4 not operated Non-surgical group: Within 30 days after randomization
Description: Only serious adverse events were assessed
Arm/Group | Surgical Group | Non-surgical Group
Serious Adverse Events (participants affected / at risk) | 14/97 | 2/98
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Group (N=97) | Non-surgical Group (N=98)
Fatal stroke (Nervous system disorders) | 1 (1) | 0 (0)
Non-fatal Stroke (Nervous system disorders) | 13 (13) | 2 (2)
Transient ischemic attack (Nervous system disorders) | 4 (4) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epidural/subdural hematoma (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Surgical site infection (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Deep venous thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation/flutter (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No